CLINICAL TRIAL: NCT03830996
Title: Weekly Plasma EBV DNA for Non-metastatic Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Victor H.F. Lee, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: WeeklyEBV
Record Dates: First submitted 2019-02-04; First posted 2019-02-05 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nasopharyngeal carcinoma (NPC) is an endemic malignancy in Southern China, Hong Kong, Taiwan, Singapore and Malaysia. It is highly associated with Epstein-Barr virus (EBV). Radiation therapy alone is indicated for early stage I to II diseases while concurrent chemoradiation is required for more advanced stage III to IVB diseases. Intensity-modulated radiation therapy (IMRT) is the standard radiation technique for NPC, in virtue of its superior target coverage and dose sparing to adjacent critical organs-at-risks.

Plasma EBV DNA and other novel plasma biomarkers have been extensively investigated in NPC. Previous studies have proven their predictive and prognostic values in NPC diagnosis, surveillance and survival outcomes.

Investigators would like to investigate the roles of plasma biomarkers including plasma EBV DNA on treatment response evaluation, survival and prognosis on NPC, in the modern era of precision radiation therapy. This will help provide important information on refining on the current edition of AJCC/UICC staging classification.

DETAILED DESCRIPTION:
Patients with histologically confirmed previously untreated NPC are be recruited to join tis study. The study has obtained approval from local institutional review board.

After written informed consent, baseline investigations including blood tests for routine hematology, biochemistry and plasma EBV DNA will be taken. Only 3ml of EDTA blood will be taken for plasma EBV DNA and other potential biomarkers. Patients will also undergo baseline imaging investigations including positron-emission tomography with integrated computed tomography (PET-CT) and magnetic resonance imaging (MRI) of the head and neck regions. An routine nasoendoscopy and nasopharyngeal biopsies will be obtained to confirm and delineate the mucosal extent of the disease.

If confirmed non-metastatic, patients will be treated with IMRT using 7-9 radiation beams. A total dose of 70Gy in 33-35 fractions over 6.5 to 7 weeks will be given. For advanced stage III to IVB diseases, concurrent chemoradiation using cisplatin 100mg/m2 on Day 1, 22 and 43 of IMRT followed by 3 cycles of adjuvant chemotherapy with cisplatin 80mg/m2 on Day 1 and 5-FU 1000mg/m2 from Day 1 to Day 4 every 4 weeks for 3 more cycles starting 4 weeks after completion of IMRT will also be given. Some patients will also receive induction chemotherapy with cisplatin100mg/m2 on Day 1 and 5-FU 1000mg/m2 on Day 1 to 5, administered every 3 weeks for 3 cycles before commencement of chemoradiation, at the discretion of treating oncologists if the primary tumours are close to critical organs e.g. brainstem, optic chiasm or optic nerves.

After treatment patients will undergo nasopharyngeal biopsies, patients will undergo nasopharyngeal biopsies again at 8 weeks after completion of IMRT to confirm histological complete local remission. Blood will be taken again on the same day for plasma EBV DNA and other potential biomarkers. Additional biopsies and salvage local treatment e.g. brachytherapy, stereotactic or IMRT boost will be offered to patients who have persistent local disease at 12 weeks after completion of IMRT. If complete local remission is confirmed, patient will have regular follow up every 3 to 4 months for surveillance and survival outcomes. Regular imaging with MRI and CT scans every 3 to 4 months will also be arranged as well. Plasma EBV DNA will be measured at weekly intervals until EBV DNA is undetectable.

For those with metastatic diseases, systemic chemotherapy (platinum-based chemotherapy) will be offered. Blood taking for plasma EBV DNA and other potential biomarkers at baseline before chemotherapy commencement and then after every 3 cycles will be arranged. Imaging examinations with CT and MRI scans will be arranged at baseline and then after 3-4 cycles of chemotherapy for tumour response evaluation.

The trend of baseline and serial plasma EBV DNA will be monitored prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed previously untreated nasopharyngeal carcinoma

Exclusion Criteria:

* Patients who are pregnant or lactating
* Patients who are not mentally capable of giving written informed consent
* Patients with performance status ECOG=3 or above or patients who are expected not able to tolerate radiation therapy and/or chemotherapy
* Patients who refuse active treatment for their nasopharyngeal carcinoma
* Patients who cannot comply with radiation therapy and/or chemotherapy for their nasopharyngeal carcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically confirmed previously untreated nasopharyngeal carcinoma (NPC) will be invited to join this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  Progression-free survival is calculated from the date of diagnosis of NPC to the date of progression of NPC or the date of death from any cause, whichever comes earlier.

SECONDARY OUTCOMES:
Overall survival | 3 years
  Overall survival is calculated from the date of diagnosis of NPC to the date of death from any cause
Distant metastasis-free survival | 3 years
  Distant metastasis-free survival is calculated from the date of diagnosis of NPC to the date of distant metastasis or date of death from any cause, whichever comes earlier.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Lee, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan SK, Chan SY, Choi HC, Tong CC, Lam KO, Kwong DL, Vardhanabhuti V, Leung TW, Luk MY, Lee AW, Lee VH. Prognostication of Half-Life Clearance of Plasma EBV DNA in Previously Untreated Non-metastatic Nasopharyngeal Carcinoma Treated With Radical Intensity-Modulated Radiation Therapy. Front Oncol. 2020 Aug 21;10:1417. doi: 10.3389/fonc.2020.01417. eCollection 2020. PMID 32974150